CLINICAL TRIAL: NCT03227978
Title: PCL (Poly-ε-caprolactone) Mesh Pleurodesis in Thoracoscopic Treatment of Primary Spontaneous Pneumothorax
Brief Title: PCL (Poly-ε-caprolactone) Mesh Pleurodesis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1060006968
Record Dates: First submitted 2017-07-11; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: PCL Pleurodesis
Keywords: pleurodesis; PCL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCL mesh group (Experimental): Intervention: The participants will be received thoracoscopic bullectomy and abrasion of pleura, then PCL mesh will be applied over the lung.
  Interventions: Combination Product: PCL mesh pleurodesis

INTERVENTIONS:
Combination Product: PCL mesh pleurodesis — Coverage of the lung surface by PCL mesh

SUMMARY:
Recent advances in thoracoscopic surgery have made it a commonly used technique for treating spontaneous pneumothoraces and preventing recurrence. The goal of surgical treatment is to find the offending bleb, remove it, and do some manipulation to encourage pleural symphysis. Methods of thoracoscopic pleural symphysis have included mechanical abrasion and instillation of chemical irritants. Each method reduces the rate of pneumothorax recurrence to a certain degree, but the recurrence rates after thoracoscopic surgery are widely varied in the literature. Although several articles show significantly lower rates, there are also articles demonstrating that the recurrence rates of pneumothorax after thoracoscopic surgery ranged between 5 and 12%, which are higher than the rates reported after open thoracotomy. It is suggested that a less intense pleural inflammatory reaction is induced by thoracoscopic procedure than by thoracotomy. Besides, post-pleurodesis severe pain and bleeding were encountered frequently. A potential alternative to increase the intensity of pleural inflammation and thereby prevent pneumothorax recurrence is film pleurodesis. Only few studies have been reported where more than one film pleurodesis has been tried, and the mechanism of film pleurodesis remains unclear.

Poly-ε-caprolactone (PCL) is a FDA-approved biomaterial with a slow degradation time of approximately 24 months when degraded by hydrolysis only. Recently, some investigators combined PCL with other biomaterials such as chitosan, polyethylene glycol, hyaluronic acid to produce anti-adhesion barrier for clinical applications. However, only few studies report PCL only could provide anti-adhesion effect. In contrast to common complications of postoperative abdominal adhesions, adhesion (or pleurodesis) is an important therapeutic tool to control the incidence of recurrent pneumothorax. We suppose that if a biomaterial induces adhesion following abdominal surgery, perhaps it may be applied to pleurodesis tool for preventing recurrence of spontaneous pneumothorax. We hypothesized that PCL membrane-induced pleurodesis can be achieved intrapleurally.

DETAILED DESCRIPTION:
Primary spontaneous pneumothorax usually occurs in young, lean young men. In most cases, the cause of pneumothorax is rupture of blebs at the apex of the lung. Traditionally, bullectomy with mechanical pleurodesis through thoracotomy is indicated in patients with recurrence or persisted air leakage. The possible causes of recurrent pneumothorax and prolonged air leakage are missed bleb surrounding the endoscopic suture line or suboptimal suturing or healing of the thoracoscopic suture. To prevent these complications, a novel method using coverage of the endoscopic suture line by a large absorbable vicryl mesh during thoracoscopic surgery was proved to be safe and feasible. Theoretically, the mesh can strengthen the suture line and induce local fibrosis surrounding the suture line, and reduce the rate of recurrent pneumothorax and prolonged air leakage. To prove this hypothesis, we will conduct a prospective randomized trial in National Taiwan University Hospital. We will enroll 10 patients with primary spontaneous pneumothorax who will be assigned to PCL mesh pleurodesis after thoracoscopic bullectomy and pleural abrasion. The primary endpoint is to check the biocompatibility of PCL mesh. The secondary endpoint is to evaluate the safety after thoracoscopic bullectomy and pleural abrasion.

ELIGIBILITY:
Inclusion Criteria:

* Primary spontaneous pneumothorax patients who require thoracoscopic bullectomy and pleurodesis

Exclusion Criteria:

* chronic obstructive pulmonary disease, hemopneumothorax, catamenial pneumothorax, pregnant, malignancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
blood pressure and temperature | three days
  mmHg and celsius degree

SECONDARY OUTCOMES:
pain scale | 3 days, 1 month and 6 months
  from 0 to 9

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shing Chen, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: Undecided